CLINICAL TRIAL: NCT03099720
Title: Role of Ropivacaine Postincisional Infiltration With Intraperitoneal Instillation Analgesia in Postoperative Pain Relief in Patients Undergoing Non Descent Vaginal Hysterectomy: Randomized Controlled Trial
Brief Title: Local Analgesia to Prevent Pain in Patient Undergoing Removal of the Uterus Through Vaginal Route
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Eman Omran, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 3777
Record Dates: First submitted 2017-03-20; First posted 2017-04-04 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Participants are given ropivacaine (0.5%) at a total dose of 50 ml, 30 ml of which is injected locally and 20 ml into the peritoneum once before the end of operation as pre-emptive analgesia.
  Interventions: Drug: Ropivacaine
- control group (Placebo Comparator): Participants are given a placebo in the form of fluid injection of saline (0.9%) at total of 50 ml, 30 ml of which is injected locally and 20 ml into the peritoneum once before the end of operation
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ropivacaine — local anesthetic will be given locally at the site of operation to decrease the level of pain after operation
  Arms: intervention group
Drug: Placebo — placebo fluid will be given at the site of operation locally
  Arms: control group

SUMMARY:
Following a hysterectomy, women tend to experience high levels of pain, and many require strong pain killers after the procedure. Ropivacaine is a local anaesthetic drug (injectable numbing medication) which works by blocking pain signals. The aim of this study is to find out whether injections of ropivacaine during surgery can help provide effective pain relief after surgery.Women aged between 45 and 70 who are having a vaginal hysterectomy can participate in the trial. Participants are randomly allocated to one of two groups. Those in the first group are given injections of ropivacaine at the site of the wound and in the peritoneum (space in the body that holds the organs in the abdomen) and those in the second group are given injections of a saline fluid in the same places that offers no pain relief before the end of their surgery. Participants in both groups are then regularly asked to rate their pain levels up to 24 hours after surgery. In addition, the pain killers they receive and length of hospital stay are recorded. There is a chance that the participants who receive the ropivacaine will benefit from lower pain levels after surgery. There are no notable risks of participating.

DETAILED DESCRIPTION:
At end of the vaginal hysterectomy operation, the gynecologist will inject the uterosacral, cardinal ligaments, adnexal areas and the vaginal edge with 15 ml of either the ropivacaine solution or the placebo fluid in each side, then 20 ml will be instilled inside the peritoneum. Analgesia will be given on request after operation. Visual analogue score of 0 to 100 mm will be used to assess the degree of pain, with 0 indicating no pain and 100 indicating worst pain.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. 45 to 70 years old
3. Scheduled for NDVH (non descent vaginal hysterectomy) for benign indications without need for oophorectomy or vaginal reconstructive surgery

Exclusion Criteria:

1. Patient weight less than 50 kg
2. Allergy to amide local anesthetic
3. Dementia or mental retardation to a degree which would interfere with data collection
4. Contraindication to non descent vaginal hysterectomy

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
pain score | At 2 hours post--operatively.
  Pain is measured by the patient using the visual analogue score

SECONDARY OUTCOMES:
Time in hours to get out of bed after operation | at 12 hours post--operatively
  Time in hours to get out of bed after operation is measured by a nurse responsible for the patient
Hospital stay in days | Up to 4 weeks post-operatively
  Hospital stay in days is measured by a nurse
Total Narcotic dose (Nalbuphine) | Up to 24 hours post--operatively
  Total Narcotic dose (Nalbuphine) is measured by a nurse
Total parenteral NSAID (diclofenac sodium) used in the first 24 hours after surgery | at 24 hours post-operatively
  Total parenteral NSAID (diclofenac sodium) used in the first 24 hours after surgery is measured by a nurse
Proportion of patients with nausea and vomiting in the first 24 hours | At 24 hours post--operatively
  Proportion of patients with nausea and vomiting in the first 24 hours is measured by a nurse
Time spent in the post-anesthesia care unit | Up to 24 hours post--operatively
  Time spent in the post-anesthesia care unit is measured by a nurse

OTHER OUTCOMES:
Pain score | At half hour post-operatively
  Pain is measured by the patient using the visual analogue score
Pain score | At one hour post-operatively
  Pain is measured by the patient using the visual analogue score
Pain score | At 4 hours post-operatively
  Pain is measured by the patient using the visual analogue score
Pain score | At 8 hours post-operatively
  Pain is measured by the patient using the visual analogue score
Pain score | At 12 hours post-operatively
  Pain is measured by the patient using the visual analogue score
Pain score | At 24 hours post-operatively
  Pain is measured by the patient using the visual analogue score

CONTACTS AND LOCATIONS:
Overall Officials: Eman Omran, M.D., Principal Investigator — Cairo University
Locations (1):
- Banha University, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided